CLINICAL TRIAL: NCT06759207
Title: Assessment of Corneal Topography and Densitometry in Rheumatoid Patients: A Prospective Case Control Study
Brief Title: Assessment of Corneal Topography and Densitometry in Rheumatoid Patients
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Elshimaa A.Mateen, Assistant Professor, Sohag University
Other Study IDs: Soh-Med-24-12-12PD
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cornea
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid arthritis patients: Pentacam

SUMMARY:
Corneal transparency is a result of its unique ultrastructure with collagen fibrils regularity, integrity of connective tissue, and balanced keratocyte components. Corneal densitometry is known to be altered in cases corneal haze or scar, but recently it is assumed to be altered earlies in presence of a systemic inflammatory disease, even before clinical manifestations take place.

The aim of this study is to assess changes in corneal topography and corneal densitometry in RA patients with clinically clear corneas and to compare these results with those of healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with rheumatoid arthritis

Exclusion Criteria:

* corneal opacity; severe dry eye; glaucoma; any inflammatory ocular disorder or infection including blepharitis, conjunctivitis, meibomitis and dacryocystitis; central or peripheral thinning evident in slit-lamp examination; history of ocular surgery, trauma, or contact lens use; and patients using any topical medication other than artificial tears will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients have RA presented for ophthalmic clinic during the period of the study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Corneal topographic changes and densitometry in patients with rheumatoid arthritis | one year

CONTACTS AND LOCATIONS:
Overall Officials: Elshimaa A.Mateen, Doctor, Principal Investigator — Assistant Professor
Locations (2):
- Egypt (2):
  - Amr Mounir, Sohag
  - Elshimaa A.Mateen, Sohag